CLINICAL TRIAL: NCT04959513
Title: Alveolar Ridge Augmentation Using GBR With L-PRF Bone Block in Early Healing Phase After Dental Extraction: a Consecutive Case Series
Brief Title: GBR With L-PRF Bone Block in Early Healing Phase After Extraction
Acronym: LPRF-GBR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Geistlich Pharma AG (Industry)
Responsible Party: Principal Investigator, Lasserre, Principal Investigator, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/19OCT/516
Record Dates: First submitted 2021-06-11; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Alveolar Ridge Augmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GBR with L-PRF bone block (Experimental): Guided bone regeneration using Leukocyte and platelet-rich fibrin
  Interventions: Procedure: LPRF bone block

INTERVENTIONS:
Procedure: LPRF bone block — Guided bone regeneration using an L-PRF bone block (composite graft composed of a xenograft, a membrane from the patient's blood and a collagenous membrane) after a short healing period of 6 to 8 weeks after tooth extraction

SUMMARY:
When the practitioners have to place an implant, it is necessary to have a sufficient amount of bone. This study propose to manage clinical situations by an approach using guided bone regeneration using an L-PRF bone block (composite graft composed of a xenograft, a membrane from the patient's blood and a collagenous membrane) after a short healing period of 6 to 8 weeks after tooth extraction. Alveolar ridge changes will be evaluated regarding soft and hard tissues up to 6 months.

DETAILED DESCRIPTION:
When the practitioners have to place an implant, it is necessary to have a sufficient amount of bone. After a tooth extraction, a bone remodeling process leads to a resorption of the various sockets components. The spontaneous healing of an extraction may result in an unsuitable site for the implant placement. It is therefore sometimes necessary to perform an alveolar ridge preservation (ARP) at the time of extraction at the future implant site to compensate for this natural resorption. However, some clinical situations don't allow ARP (infection, significant bone loss, etc.) at the time of extraction. In these situations where alveolar preservation is not indicated and bone augmentation is required to recover or preserve correct bone anatomy for implant placement, other techniques must be used. Thus, in this study, the investigators propose to manage these clinical situations by an approach using guided bone regeneration using an L-PRF bone block (composite graft composed of a xenograft, a membrane from the patient's blood and a collagenous membrane) after a short healing period of 6 to 8 weeks after tooth extraction. This early approach allows soft tissue healing (easier primary closure to cover the graft), take advantage of the residual bone architecture of the socket (only at the beginning of its resorption) and allows infection resorption at the extraction site.

The outcomes are the volumetric changes of the soft and hard tissue. To evaluate this volumetric changes, 3 CBCTs and 3 digital impressions will be made at 3 different times: before extraction, before guided bone regeneration and before implant placement (5 to 8 months after regeneration).

Patients will be recruited at Cliniques Universitaires Saint-Luc, participation will be voluntary without any obligation. To be included in the experiment, patients will have to have at least one tooth from the antero-superior sector that must be extracted with the need for pre-implant bone regeneration. This need for guided bone regeneration will be based on a three-dimensional radiological examination.

The chronology of the experiment is :

1. First consultation to make the diagnosis, explain the experiment and sign the informed consent.
2. 1st CBCT (Cone Beam Computed Tomography) and 1st digital impression.
3. Surgery: extraction of tooth(s).
4. 2nd CBCT, digital impression and control of the healing of the extraction site 10 to 15 days after extraction.
5. Surgery: Guided bone regeneration 6 to 8 weeks after extraction.
6. Control of the healing of the site 10 to 14 days after regeneration.
7. 3rd CBCT, 3rd digital impression 5 to 8 months after regeneration.
8. Surgery: Implant placement. The data analysis will be done clinically with control visits after the different surgeries and volumetrically with CBCTs and optical impressions. The impressions and the radiographic images will be analysed used dedicated application (MeVisLab for the CBCTs and Gom Inspect for the impressions).

ELIGIBILITY:
Inclusion Criteria:

* To be over 18 years old.
* Be in good general health.
* Have at least one monoradicular tooth (premolar, canine or incisor) that must be extracted with the need for bone regeneration and one or more implants afterwards.
* Have a DPSI (Dutch Periodontal Screening Index) ≤ 2.

Exclusion Criteria:

* Being a smoker.
* Have "active" periodontal problems, have a DPSI > 2.
* Have a contraindication to the insertion of an implant and/or oral surgery.
* Have an active inflammatory and/or autoimmune disease of the oral cavity.
* Treatment with immunosuppressants, corticosteroids or biphosphonates.
* Have a history of cancer, radiotherapy or chemotherapy for cancer within the last 5 years.
* Have insulin-dependent diabetes.
* Have a blood disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Gain in ridge width in millimeters | 5 to 8 month after guided bone regeneration
  Volumetric analysis of hard tissue using CBCT. They will be performed before extraction (T0), before guided bone regeneration (T1) and 6 months after regeneration before implant placement (T2). The CBCT done at T0 will be used as a reference for comparison with the CBCT T1 and T2. A high-resolution scanning protocol will be used with fixed exposure parameters and the CBCT will be adjusted to the target area to allow a significant reduction in irradiation dose. The DICOMs (Digital Imaging and Communication in Medicine) will be analysed using a dedicated application. The images taken at different times will be superimposed with an automatic algorithm and compared by 2D and 3D volumetric measurements.

SECONDARY OUTCOMES:
Volumetric changes of the soft tissue in millimeters | 5 to 8 month after guided bone regeneration
  Volumetric analysis of soft tissue using digital impressions. They will be made before extraction (T0), before guided bone regeneration (T1) and 6 months after regeneration before implant placement (T2). The impressions taken at the different times will be compared in analysis software. Oral-lingual or oral-palatal measurements will be taken in the center of the edentulous site at 1mm, 3mm and 5mm from the gingiva.
Need or not of an additional grafting procedure (yes or no) | 5 to 8 month after guided bone regeneration
  Analyse of the need for further regeneration before the implant is placed.
Analysis of the implant's osseointegration (ISQ) | up to 12 months
  An analysis of the osseointegration of the implant using a dedicated device (Osstell IDx, Osstell AB, Göteborg, Sweden).
Patient reported outcomes mesures (VAS Scale) | through study completion, an average of 1 year
  Analysis of the patient's feeling thanks to a "Visual Analog Scale" scale carried out 1 week after the regeneration surgery.
Occurrence of an adverse effect | through study completion, an average of 1 year
  Analysis of the infection rate after regeneration.

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Lasserre, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Clinique Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No